CLINICAL TRIAL: NCT00598299
Title: Department of Ophthalmology, National Taiwan University Hospital
Brief Title: Comparison of the Effects on Promoting Corneal Epithelial Wound Healing Between Human Auto-Serum and Cord Blood Serum
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wei-Li Chen, Department of Ophthalmology, National Taiwan University Hospital
Other Study IDs: 20072037R
Record Dates: First submitted 2008-01-10; First posted 2008-01-21 (Estimated); Last update posted 2008-11-04 (Estimated); Status verified 2008-10

CONDITIONS: Eye Injuries
Keywords: corneal epithelium
MeSH Terms: conditions — Eye Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A: Healthy adult serum
  Interventions: Procedure: venous puncture; Other: obtain serum from perripheral blood or cord blood
- B: cord blood serum
  Interventions: Procedure: venous puncture; Other: obtain serum from perripheral blood or cord blood

INTERVENTIONS:
Procedure: venous puncture — venous puncture
Other: obtain serum from perripheral blood or cord blood — obtain serum from perripheral blood or cord blood

SUMMARY:
Human serum eye drops have been successfully used in the treatment of severe ocular surface disorders and the enhancement of corneal wound healing. Umbilical cord serum is also proven to be effective in treatment of dry eye and persistent corneal epithelial defects. However, there are limited studies comparing the corneal epithelial wound healing promoting effects between these two blood derived products. The purpose of this study is to test the corneal epithelial wound healing promoting effects between auto serum and human cord blood serum. Primary cultured bovine corneal epithelial cells were used as the model to investigate wound healing, cell proliferation and migration by means of scratch corneal wound healing assay evaluation, MTS assay and Boyden chamber migration assay in response to human serum and umbilical cord serum. The concentrations of EGF, TGF-β1, and fibronectin were also compared between human serum and umbilical cord serum with ELISA kits.

DETAILED DESCRIPTION:
Human serum eye drops have been successfully used clinically in the treatment of severe ocular surface disorders and the enhancement of corneal wound healing. Umbilical cord serum is also proven to be effective in treatment of dry eye and persistent corneal epithelial defects. However, there are limited studies comparing the corneal epithelial wound healing promoting effects between these two blood derived products. The purpose of this study is to test the corneal epithelial wound healing promoting effects between auto serum and human cord blood serum. Primary cultured bovine corneal epithelial cells were used as the model to investigate wound healing, cell proliferation and migration by means of scratch corneal wound healing assay evaluation, MTS assay and Boyden chamber migration assay in response to human serum and umbilical cord serum. The concentrations of EGF, TGF-β1, and fibronectin were also compared between human serum and umbilical cord serum with ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

healthy volunteers

Exclusion Criteria:

unhealthy volunteers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: heahty adult volunteers and donated cord blood
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-04; Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fung-Rong Hu, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan